CLINICAL TRIAL: NCT06356207
Title: NeuroArrhythmias Area Registry of AIAC (NAARA) Syncope-Asystole Latency Time in Tilt Table Test (SALT-TILT) Study
Brief Title: Syncope-Asystole Latency Time in Tilt Table Test: The SALT-TILT Study
Acronym: SALT-TILT
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Bolzano (Other)
Responsible Party: Principal Investigator, Matthias Unterhuber, Principal Investigator, Azienda Ospedaliera di Bolzano
Other Study IDs: 113-2023
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Syncope; Pacemaker; Asystole; Neurally Mediated Syncope
Keywords: Syncope; Pacemaker; Tilt Table Test; Asystole; SALT; Syncope-Asystole Latency Time
MeSH Terms: conditions — Syncope; Heart Arrest; Syncope, Vasovagal | interventions — Tilt-Table Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by neuronally mediated syncope
  Interventions: Diagnostic Test: Tilt Table Test

INTERVENTIONS:
Diagnostic Test: Tilt Table Test — The main goal of the study is to evaluate the time elapsed between the T-LOC during Video Tilt Table Testing and the asystole at the ECG using a national registry and to assess its predictive value in patients undergoing invasive treatment. The hypothesis is that a vasodepressive component could lessen the effect of pacing in a patient, leading to cerebral hypoperfusion and syncope despite maintaining a stable rhythm.

SUMMARY:
Syncope is a common presenting condition. Pacemaker implantation can significantly reduce syncope recurrences in reflex syncope. However, despite careful selection, a substantial proportion of patients treated with pacemakers suffer recurrences of syncope. It is thought that a pronounced vasodepressor component may hinder the efficacy of pacing in patients, preventing adequate cerebral perfusion during the reflex, thus relativizing the anti-bradycardia function of the pacemaker to prevent syncope. It is hypothesised that the time elapsed from the actual loss of consciousness to the asystole recorded on the ECG during Tilt Table Test may be predictive in terms of response to pacemaker therapy, so this parameter becomes the subject of the present study.

DETAILED DESCRIPTION:
Syncope is a common leading affection and is responsible for 1-3% of the presentations in emergency departments and up to 3% of inpatient admissions. Syncope poses often a diagnostic and therapeutic challenge for the attending physician and is often misdiagnosed or underdiagnosed. Patients can be treated with pacemaker implantation when the syncope cause is a cardioinhibition with documented asystole during the syncopal event. When accurately selected, patients benefit from pacemaker therapy with a significant reduction of syncope recurrence in the follow up. However, a substantial portion of the patients (approx. 25%) experience recurrence of syncope despite optimal pacemaker therapy. The underlying mechanism is not well understood and object of the current study.

The main target of the study is to evaluate the time elapsed between the T-LOC during Video Tilt Table Testing and the asystole at the ECG using a registry and to assess its predictive value in patients undergoing invasive treatment. The hypothesis is that a vasodepressive component could lessen the effect of pacing in a patient, leading to cerebral hypoperfusion and syncope despite maintaining a stable rhythm.

This is a prospective, multi-center observational study with 2 year follow-up of patients. Patients eligible for invasive treatment of reflex syncope are included.

If after guideline-directed implantable loop recorder insertion no cardioinhibition has been recorded, the patient is included automatically in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for invasive treatment according to the ESC Guidelines for pacing 2021
* Written informed consent

Exclusion Criteria:

* Other condition which explains syncope cause other than reflex syncope
* Structural heart disease (valvular, ischaemic, cardiomyopathies)
* Pregnancy
* Patient denial to be recorded on video during tilt table test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by neurally mediated syncope eligible for invasive treatment according to the ESC Guidelines for pacing 2021
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
SALT (Syncope-Asystole Latency Time) | From enrollment to end of treatment 2 weeks
  • Syncope to asystole latency time (SALT) and its prognostic value regarding freedom of syncope recurrence after pacemaker implantation

SECONDARY OUTCOMES:
Recurrence of syncope | From enrollment to treatment end 24 months
  • Recurrence of syncope in patients treated with different pacemaker configurations (DDD-CLS, DDD-RDR, DDDrr) and Neurocardioablation
Recurrence of syncope | 24 months
  • Recurrences of syncope in treated patients selected by CSM or loop recorder and negative or positive vasodepressive VTTT

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria di Bolzano, Bolzano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT06356207/Prot_SAP_000.pdf